CLINICAL TRIAL: NCT04782011
Title: Feasibility of Using the Chemical Classification System/Defined Daily Doses Tool to Monitor Antibiotic Use at Primary Healthcare Facilities in Southwestern Uganda
Brief Title: Using the ATC/DDD to Monitor Antibiotic Use at Lower Primary Care Facilities in Southwestern Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBS-HDREC-564
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: ATC/DDD; Antibiotic Utilization
Keywords: ATC/DDD; Antibiotic utilization; Lower primary care facilities; Southwestern Uganda

STUDY DESIGN:
Intervention Model Description: The number of health facilities will be split evenly between the intervention and non intervention arms. These will be randomly selected in the districts of Mbarara, Bushenyi and Kasese.
Masking Description: Being a feasibility study that will use patient records, no blinding will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATC/DDD arm (Experimental): The intervention is the introduction of the ATC/DDD including the training of healthcare workers on its importance and usage in monitoring antibiotic use. The unit of intervention will be a health facility. Antibiotic prescriptions and antibiotic utilization records for adult patients (in-patients and ambulatory) from the selected facilities will be enrolled in the study.
  Interventions: Behavioral: ATC/DDD
- Control arm (No Intervention): The health care workers will continue with standard practice. However, the research team will collect data on antibiotic prescriptions and antibiotic utilization for adult patients (in-patients and ambulatory) from the selected facilities. The data will be compared with that of the intervention arm.

INTERVENTIONS:
Behavioral: ATC/DDD — The intervention is the introduction of the ATC/DDD including the training on its importance and usage in monitoring antibiotic use at a given primary care facility.
  Arms: ATC/DDD arm

SUMMARY:
This is a non blinded two arm cluster randomized control trial, aimed at assessing the feasibility of using the Anatomical Therapeutic Chemical Classification/define Daily Doses system tool to monitor antibiotic use at lower primary levels of care in Uganda.

DETAILED DESCRIPTION:
The study will evaluate the feasibility of using the ATC/DDD in three districts of Southwestern Uganda. The unit of intervention will be a health facility. Eighteen (18) randomly selected government owned health facilities at levels II, III and IV will be split evenly between the intervention and non intervention arms. Antibiotic prescriptions of new adult (in-patients and ambulatory) patients with antibiotic utilization records from the selected facilities will be enrolled in the study. The intervention is the introduction of the ATC/DDD plus the training on its importance and use by healthcare providers. The facilities selected will be far apart from each other to avoid contamination.

Intervention arm: The ATC/DDD tool shall be piloted in all selected facilities of the 3 randomly selected districts of Mbarara, Bushenyi and Kasese. The prescribers at these facilities will be trained about the importance and usability of the ATC/DDD tool. A pre and post assessment of the prescribers understanding of the tool's usability will be done prior to piloting the tool. This will guide the focus of the training and any other necessary support after the training. The trained prescribers will use the latest tool version to evaluate drug utilization of antibiotics (anti-infectives for systemic use) used at their respective facility levels for a period of 6 months. Prescriptions and drug administration reviews will be done in three phases and for 5 days following the National Medical Stores delivery schedule for medicines, that is, shortly after delivery of drugs (phase 1), midway (phase 2) and towards the end of the delivery period (phase 3). The evaluation will involve computation of antibiotic utilization parameters using the latest version of the ATC/DDD by both the trained healthcare providers and an independent research team. Findings will be compared for both groups to ensure implementation infidelity. .

Patients and antibiotic utilization records:

1. For inpatients: On the day of patient recruitment, health workers will routinely conduct baseline assessment of the consented patients to obtain data on demographics, clinical conditions and medications. Daily reviews of patients shall be conducted as routinely done by the clinicians until discharge, referral, death or loss to follow-up. A data extraction template will then be used to capture both baseline and daily follow-up patient information . Medication data will be obtained from the patient's hospital file (clinical notes, treatment sheets and drug administration charts), dispensing records of ward units, pill count validation of a patient's oral medication (capsules, tablets,) and of unused injectable medicine vials or ampoules in the possession of the patient or the caregiver. This will be done on a daily basis.
2. For ambulatory patients: Only prescription data will be obtained from Out-patient Department (OPD) registers, dispensing logs and/or patients' charts using a data extraction template.

Non-intervention arm: These will continue with the standard practice. However, the research team will collect data during the respective phases highlighted in the intervention arm for computation using the latest version of the ATC/DDD tool and comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Health facility: The facility will be government owned that receives antibiotics from National Medical Stores using the current schedule and has no ongoing antibiotic use related intervention study.
2. Prescribers: Male and female prescribers at primary care facilities in the selected districts of Mbarara, Bushenyi and Kasese will be recruited. Prescribers with an experience of at least 3 months in antibiotic prescribing and inventory at these facilities will be included in the study. These shall be identified through the in-charges of the respective facilities.
3. Patients: New male and female adult patients (18 years and above) receiving antibiotic medication will be enrolled.
4. Antibiotic utilization records: Antibiotic prescriptions and administration charts for new patients at selected health facilities.

Exclusion Criteria:

1. Patients: Those who are too sick to cooperate
2. Prescriptions: Ineligible prescriptions and the prescriber cannot be reached for clarifications.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1406 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Trends in antibiotic utilization for both the intervention and non intervention arms | 3 months
  Computation of antibiotic utilization parameters across the different facility levels will be done using the latest version of the ATC/DDD tool. Antibiotic use by clinical condition data will be analyzed using working diagnoses that will be classified into diagnostic groups using the latest version of the International Classification of Diseases, Clinical Modification (ICD-10-CM) diagnosis codes as a guide. Findings of both arms will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Mukonzo, PhD, Study Director — Makerere University; Vincent Batwala, PhD, Study Director — Mbarara University of Science and Technology
Locations (1):
- Hanifah Nantongo, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
I do not intend to share the data